CLINICAL TRIAL: NCT05999487
Title: Dobutamine Versus Milrinone in Management of Critically Ill Low Cardiac Output Pediatric Patients at Cairo University Children's Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Gamal, pediatric resident, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: inotropes in pediatrics
Record Dates: First submitted 2023-05-05; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Dobutamine, Milrinone , Pediatrics , Low Cardiac Output
MeSH Terms: conditions — Cardiac Output, Low | interventions — Dobutamine; Milrinone

STUDY DESIGN:
Who Masked: Investigator
Masking Description: . Cardiac assessment will be done by a blinded pediatric cardiologist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients who will recieve dobutrex (Active Comparator): patient presenting with acute heart failure , who will recieve dobutrex as a result of their randomixation , startng dose will be 5 mic , assesing their need for tittration of dose , the need for addition of another inotrope , the prescence of any side effects and the duration of inotropic use for reaching hemodynamically stable state
  Interventions: Drug: Dobutamine
- patients who will recieve milirinone (Experimental): patient presenting with acute heart failure , who will recieve milirinone as a result of their randomixation , startng dose will be 0.25 mic , assesing their need for tittration of dose , the need for addition of another inotrope , the prescence of any side effects and the duration of inotropic use for reaching hemodynamically stable state
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Patient randomization will be done by a computer based generation , serial enveloped numbers will be taken for the patients. Cardiac assessment will be done by a blinded pediatric cardiologist. If at any time the randomly assigned therapy considered to be failed or unsafe to continue, the treating physician will discontinue randomization and will continue with the appropriate medication according to the patients need.
  Milrinone will start by 0.25 , 0.5 , 0.75 we can titrate up with time interval 3 hours after re-assessment.
  Dobutamine will start by 5, 10 , 15, 20 we can titrate with time interval 15 mins after re-assesment.
  Other Names: milrinone

SUMMARY:
The aim of the study is to detect wither dobutamine or milrinone have a privilege in the management of low cardiac output pediatric patients over the other.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) enrolling critically ill patients with low cardiac output syndrome (LCOS) admitted at pediatrics emergency and intensive care units ,Cairo University Children's Hospital, identified by treating medical team as requiring initiation of inotropic therapy based on healthcare team assessment of :

* Capillary refill time > 3 sec
* Hypotension (less than the 5th percentile or less than 90/50 mmHg for children 10 years or older (Kleinman et al.,2010) (Haque et al .,2007)
* Oliguria (urine output that is less than 1 mL/kg/h in infants, less than 0.5 mL/kg/h in children ) (Nakano et al.,2022)
* Metabolic acidosis with base excess > -2 (Nakano et al.,2020)

Patient randomization will be done by a computer based generation , serial enveloped numbers will be taken for the patients. Cardiac assessment will be done by a blinded pediatric cardiologist. If at any time the randomly assigned therapy considered to be failed or unsafe to continue, the treating physician will discontinue randomization and will continue with the appropriate medication according to the patients need.

Every patient will be evaluated after the first 24 hours of starting the inotropic therapy by :

* pre and post inotropic therapy ICON measurements ( evaluating cardiac index and systemic vascular resistance pre and post inotropic support)
* pre and post inotropic therapy echocardiography ( evaluating systolic and diastolic dysfunction by M-mode and two dimensional methods) through measuring LV EDD cm, LV ESD cm, LV EDV ml, LVESV ml, FS% , LV mass, EF% , MAPSE cm, TAPSE cm.
* pre and post inotropic therapy clinical assessment of vital signs (heart rate , blood pressure, capillary refill time and urine output as mention before)
* The need of titration up of inotropes :

Milrinone will start by 0.25 , 0.5 , 0.75 we can titrate up with time interval 3 hours after re-assessment.

Dobutamine will start by 5, 10 , 15, 20 we can titrate with time interval 15 mins after re-assesment.

-Time to achievement of therapeutic endpoints for hemodynamics

* adequate blood pressure
* clinically adequate cardiac output ( capillary refill time < 2sec , urine output that is more than 1 mL/kg/h in infants, more than 0.5 mL/kg/h in children, full conscious )

Data will be collected for each patient in form of [ Time Frame: Through first 24 hours up to first week since admission ] :

1. Total time on inotropes (in hours)
2. Non-invasive or invasive mechanical ventilation Total number of days requiring non-invasive or invasive mechanical ventilation
3. Change in cardiac index ([CI] measured with ICON
4. Change in systemic vascular resistance [SVR] measured with ICON
5. Presence of acute kidney injury (defined as an increase in serum creatinine or a decrease in urine output or both over hours to days.) (Jacob J et al.,2020)
6. Absence of metabolic acidosis (BE -2 to 2)
7. Arrhythmia requiring medical team intervention, either through electrical or chemical cardioversion or any intravenous anti-arrhythmia medication administration
8. Need for up-titration or addition of new vasopressor therapy

ELIGIBILITY:
Inclusion Criteria:

* 1-Patients from age of 1 month to 14 years old of both sexes.

  2-Patients presenting with fluid refractory shock with low cardiac output state, evidenced by sustained hypotension (systolic blood pressure below 5th percentile for age) and end organ dysfunction (altered level of consciousness, renal or hepatic dysfunction)

  3-Clinical evidence of systemic and/or pulmonary congestion despite use of vasodilators and/or diuretics

  4-Refractory heart failure requiring admission for inotropic support.

Exclusion Criteria:

1-All other causes of pediatric shock not in need for inotropic support (eg.isolated hypovolemic shock, anaphylaxis,….)

2 - patients not fit for randomization needing specific line of management (eg. Sever hypotension patients with good filling pressure unfit for milrinone , patients previously known having sever pulmonary hypertension not fit for dobutamine ,…)

3-post cardiac surgery patients with low cardiac output manifestation.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
time to achievemnets of theraputeic endpoints of hemodynamics | first 24 hrs
  ( normal blood pressure and clinically adequate cardiac output)

SECONDARY OUTCOMES:
Correlation between the used inotropic support and the survival to discharge . | first week
Total time on inotropes and average length of stay at a pediatric intensive care unit. | first week
Need for up-titration or addition of other inotropic support. | first 24 hrs
Frequency of arrythmias and side effects encountered with the use of inotropic support in pediatrics population. | first 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Children'S Hospital, Giza, Egypt

REFERENCES:
- [Background] Haque IU, Zaritsky AL. Analysis of the evidence for the lower limit of systolic and mean arterial pressure in children. Pediatr Crit Care Med. 2007 Mar;8(2):138-44. doi: 10.1097/01.PCC.0000257039.32593.DC. PMID 17273118
- [Background] Jacob J, Dannenhoffer J, Rutter A. Acute Kidney Injury. Prim Care. 2020 Dec;47(4):571-584. doi: 10.1016/j.pop.2020.08.008. Epub 2020 Oct 1. PMID 33121629
- [Background] Jentzer JC, Coons JC, Link CB, Schmidhofer M. Pharmacotherapy update on the use of vasopressors and inotropes in the intensive care unit. J Cardiovasc Pharmacol Ther. 2015 May;20(3):249-60. doi: 10.1177/1074248414559838. Epub 2014 Nov 28. PMID 25432872
- [Background] Kleinman ME, Chameides L, Schexnayder SM, Samson RA, Hazinski MF, Atkins DL, Berg MD, de Caen AR, Fink EL, Freid EB, Hickey RW, Marino BS, Nadkarni VM, Proctor LT, Qureshi FA, Sartorelli K, Topjian A, van der Jagt EW, Zaritsky AL; American Heart Association. Pediatric advanced life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Pediatrics. 2010 Nov;126(5):e1361-99. doi: 10.1542/peds.2010-2972D. Epub 2010 Oct 18. No abstract available. PMID 20956434
- [Background] Lewis TC, Aberle C, Altshuler D, Piper GL, Papadopoulos J. Comparative Effectiveness and Safety Between Milrinone or Dobutamine as Initial Inotrope Therapy in Cardiogenic Shock. J Cardiovasc Pharmacol Ther. 2019 Mar;24(2):130-138. doi: 10.1177/1074248418797357. Epub 2018 Sep 2. PMID 30175599
- [Background] Mathew R, Di Santo P, Jung RG, Marbach JA, Hutson J, Simard T, Ramirez FD, Harnett DT, Merdad A, Almufleh A, Weng W, Abdel-Razek O, Fernando SM, Kyeremanteng K, Bernick J, Wells GA, Chan V, Froeschl M, Labinaz M, Le May MR, Russo JJ, Hibbert B. Milrinone as Compared with Dobutamine in the Treatment of Cardiogenic Shock. N Engl J Med. 2021 Aug 5;385(6):516-525. doi: 10.1056/NEJMoa2026845. PMID 34347952
- [Background] Masse L, Antonacci M. Low cardiac output syndrome: identification and management. Crit Care Nurs Clin North Am. 2005 Dec;17(4):375-83, x. doi: 10.1016/j.ccell.2005.07.005. PMID 16344207
- [Background] Nakano H, Nagai T, Honda Y, Honda S, Iwakami N, Matsumoto C, Asaumi Y, Aiba T, Noguchi T, Kusano K, Yokoyama H, Ogawa H, Yasuda S, Chikamori T, Anzai T. Prognostic value of base excess as indicator of acid-base balance in acute heart failure. Eur Heart J Acute Cardiovasc Care. 2020 Aug;9(5):399-405. doi: 10.1177/2048872619898781. Epub 2020 Jan 23. PMID 31970993
- [Background] Nakano H. Oliguria. https://emedicine.medscape.com/article/983156-overview. Updated: Feb 28, 2022. Accessed at 15-12-2022.
- [Background] Uhlig K, Efremov L, Tongers J, Frantz S, Mikolajczyk R, Sedding D, Schumann J. Inotropic agents and vasodilator strategies for the treatment of cardiogenic shock or low cardiac output syndrome. Cochrane Database Syst Rev. 2020 Nov 5;11(11):CD009669. doi: 10.1002/14651858.CD009669.pub4. PMID 33152122